CLINICAL TRIAL: NCT02952989
Title: A Phase 1, Multicenter, Open-label, Dose-escalation Study of SGN-2FF in Patients With Advanced Solid Tumors
Brief Title: A Safety Study of SGN-2FF for Patients With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to overall benefit/risk profile
Sponsor: Seagen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SGN2FF-001
Record Dates: First submitted 2016-10-27; First posted 2016-11-02 (Estimated); Last update posted 2019-07-19 (Actual); Status verified 2019-07

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Carcinoma, Renal Cell; Breast Neoplasms; Urinary Bladder Neoplasm; Carcinoma, Squamous Cell of Head and Neck; Colorectal Neoplasms; Gastric Adenocarcinoma; Gastroesophageal Junction Adenocarcinoma
Keywords: MSI-high; dMMR; PD-L1
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma, Renal Cell; Breast Neoplasms; Urinary Bladder Neoplasms; Squamous Cell Carcinoma of Head and Neck; Colorectal Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SGN-2FF (Experimental): Dose escalation and dose expansion
  Interventions: Drug: SGN-2FF
- SGN-2FF and Pembrolizumab (Experimental): Dose escalation and dose expansion
  Interventions: Drug: SGN-2FF; Drug: pembrolizumab

INTERVENTIONS:
Drug: SGN-2FF — SGN-2FF oral daily dosing.
  Other Names: 2-fluorofucose
Drug: pembrolizumab — 200 mg every 3 weeks by IV infusion
  Other Names: Keytruda
  Arms: SGN-2FF and Pembrolizumab

SUMMARY:
This study is being done to find out the side effects (unwanted effects) that are caused in patients with cancers who are given SGN-2FF. This study will also attempt to find the most suitable dose in the disease or condition being studied and look at other effects of SGN2FF, including its effect on cancer.

This study has several different parts. Part A will try to find the highest safe dose. Part B will enroll more patients to be treated at the highest safe dose or a lower dose to better understand how well SGN-2FF is tolerated. Part C will try to find the highest safe dose of SGN-2FF when it is given combined with pembrolizumab. Pembrolizumab is a standard treatment for cancer. Part D will enroll more patients to be treated at the highest safe dose of SGN-2FF combined with pembrolizumab or a lower dose of SGN-2FF to better understand how well SGN-2FF is tolerated when it is given with pembrolizumab.

DETAILED DESCRIPTION:
This is a phase 1, open-label, multicenter, dose escalation study that will examine the safety profile of SGN-2FF given orally to patients with advanced solid tumors. The primary goal of the study is to identify the maximum tolerated dose (MTD), or optimal biological dose (OBD) that does not exceed the MTD. The pharmacokinetics (PK) and antitumor activity of SGN-2FF will also be evaluated. In this study, SGN-2FF will be evaluated as monotherapy and as combination therapy with the standard approved dose of pembrolizumab.

The monotherapy portion of the study will be conducted in 2 sequential parts (Part A and Part B). Part A will enroll patients for dose escalation to estimate the MTD /OBD and help determine the dosing regimen that will be tested in Part B. The OBD will be evaluated by assessing the activity of SGN-2FF, including pharmacodynamics, PK, and other observations in dose escalation. Part B will explore the recommended dose/regimen in up to 3 focused expansion cohorts.

The combination therapy portion of the study will be conducted in 2 sequential parts (Part C and Part D). SGN-2FF will be administered orally according to the dose and schedule assigned, with a lead-in period of 2 weeks prior to pembrolizumab administration. The lead-in period may be discontinued based on emerging nonclinical and/or clinical data. Part C will enroll patients for dose escalation to estimate the MTD /OBD and the dosing regimen that will be tested in Part D. Part D will explore the recommended dose/regimen in up to 3 focused expansion cohorts.

Safety will be monitored throughout the trial by the safety monitoring committee which will meet frequently to review the emerging safety data and make dose-escalation and dosing-interval recommendations. Antitumor activity will be assessed by radiographic imaging. Patients may continue treatment until progression of their disease or intolerable side effects.

Retreatment with SGN-2FF monotherapy or with SGN-2FF and pembrolizumab combination therapy is permitted with medical monitor approval for patients who achieve stable disease, a complete response, or partial response on study and then experience disease progression after discontinuing prior treatment with SGN 2FF.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically or cytologically-confirmed, locally advanced, or metastatic solid malignancy that is relapsed, refractory, or progressing following at least 1 prior systemic therapy (Part A)
* Measurable disease by computed tomography (CT) or magnetic resonance imaging (MRI) as defined by RECIST 1.1
* Eastern Cooperative Oncology Group (ECOG) performance status of less than or equal to 1
* Patients in Part B must have histologically or cytologically-confirmed, locally-advanced, or metastatic solid malignancy within the disease indications of Part A
* Adequate baseline hematologic, renal, and hepatic function
* Patients for whom there is no further standard therapy available at the time of enrollment (Part A)
* Patients with a histologically-confirmed, advanced solid malignancy meeting one of the following criteria: (1) indication for which pembrolizumab is approved or (2) relapsed, refractory, or progressive disease following at least 1 prior therapy and for which no further standard therapy is a available (Parts C and D)

Exclusion Criteria:

* Patients with carcinomatous meningitis or active central nervous system (CNS) metastases
* Patients with recent (within 14 days) or serious ongoing infection
* Patients requiring systemic treatment with corticosteroids (greater than 10 mg prednisone equivalents) or immunosuppressive medications within 14 days of enrollment
* Patients with active known or suspected autoimmune disease or significant autoimmune-related toxicity from prior immuno-oncology therapy
* Known active or latent tuberculosis
* Uncontrolled diabetes mellitus
* History of interstitial lung disease
* Gastrointestinal abnormality that would affect absorption of SGN-2FF
* Patients tested positive for hepatitis B or with a known, active hepatitis C infection
* Women who are pregnant or breastfeeding
* Patients with deep vein thrombosis (DVT)
* Contraindication to prophylactic anticoagulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2017-02-23 (Actual); Primary Completion 2019-06-24 (Actual); Study Completion 2019-06-24 (Actual)

PRIMARY OUTCOMES:
The number of participants with adverse events that are related to treatment | Up to 90 days following last dose
  The number of patients who have side effects that are related to the study drug
The number of participants with laboratory abnormalities that are related to treatment | Up to 90 days following last dose
  The number of patients who have laboratory test results that are outside the normal range
Incidence of dose-limiting toxicities (DLTs) | 28 days from first dose
  The rate of occurrence of side effects that prevent giving more of the treatment

SECONDARY OUTCOMES:
Pharmacokinetic assessments | Relative to most recent dosing event
  Selected PK parameters, including area under the curve, maximum observed concentration, time to maximum observed concentration, and trough concentration.
Markers of fucosylation status | Up to 90 days following last dose
  Changes in pharmacodynamic biomarkers of fucosylation across dose levels
Objective response rate | Up to 90 days following last dose
  The proportion of patients who achieve a complete response (CR) or partial response (PR).
Disease control rate | Up to approximately 5 years
  The proportion of patients who achieve either complete response (CR), partial response (PR), or stable disease (SD)
Duration of response | Up to approximately 5 years
  The time from the first documentation of objective response (CR or PR) to the first documentation of tumor progression (progressive disease per response criteria or clinical disease progression) or to death due to any cause, whichever comes first
Clinical benefit rate | Up to approximately 5 years
  The proportion of patients who achieve either complete response (CR), partial response (PR), or stable disease (SD) for at least 24 weeks
Progression-free survival | Up to approximately 5 years
  The time from start of study treatment to the first documentation of tumor progression (progressive disease per response criteria or clinical disease progression) or death due to any cause, whichever comes first
Overall survival | Up to approximately 5 years
  The time from start of study treatment to date of death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: Christina Derleth, MD, Study Director — Seagen Inc.
Locations (11):
- United States (11):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - City of Hope National Medical Center, Duarte, California
  - University of Colorado Hospital / University of Colorado, Aurora, Colorado
  - Winship Cancer Institute / Emory University School of Medicine, Atlanta, Georgia
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Institute / Wayne State University, Detroit, Michigan
  - Duke University Medical Center, Durham, North Carolina
  - Providence Portland Medical Center, Portland, Oregon
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - MD Anderson Cancer Center / University of Texas, Houston, Texas
  - Seattle Cancer Care Alliance / University of Washington, Seattle, Washington